CLINICAL TRIAL: NCT01473576
Title: The Impact of Dietary Nitrate Ingestion on Muscle Protein Synthesis in Elderly Type II Diabetics
Brief Title: Impact of Nitrate Ingestion on Protein Synthesis
Acronym: PRO-Nitrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 11-3-057
Record Dates: First submitted 2011-11-03; First posted 2011-11-17 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2012-10

CONDITIONS: Muscle Protein Synthesis
Keywords: type II diabetes; protein synthesis; nitrate; elderly
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nitrates; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate (Experimental): Sodium nitrate ingestion prior to ingesting intrinsically labeled protein
  Interventions: Dietary Supplement: Nitrate
- Sodium chloride (Placebo Comparator): Sodium chloride placebo group
  Interventions: Dietary Supplement: Sodium chloride

INTERVENTIONS:
Dietary Supplement: Nitrate — 0.15 mmol/kg body weight sodium nitrate (dissolved in 250 mL water)
  Arms: Nitrate
Dietary Supplement: Sodium chloride — 0.15 mmol sodium chloride dissolved in 250 mL water.
  Arms: Sodium chloride

SUMMARY:
A diet rich in leafy green vegetables has been shown to reduce the risk of developing chronic metabolic disease. The health benefits from these particular vegetables may be attributed to their high nitrate content. Recent work suggests that dietary nitrate triggers endogenous nitric oxide release, thereby stimulating vasodilation and improving muscle perfusion in an insulin-independent manner. We hypothesize that in an insulin-resistant state, nitrate co-ingestion will increase muscle perfusion, thereby improving post-prandial delivery of nutrients to skeletal muscle tissue. Specifically, a more efficient delivery of food derived amino acids will stimulate post-prandial muscle protein synthesis and, as such, compensate for a blunted muscle protein synthetic response to food intake in the elderly. This proposal will investigate the efficacy of nitrate co-ingestion as a means to augment muscle protein synthesis in elderly, type 2 diabetes patients and may lead to a novel therapy in the clinical care of type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 70-85 years
* BMI < 30 kg/m2
* Non insulin-dependent diabetes mellitus type 2 patients (T2DM) ( >1 y since diagnoses)

Exclusion Criteria:

* Smoking
* Hypertension (according to WHO criteria)[29] and/or cardiovascular disease treated with medication containing nitrates and/or having vasodilatory effects
* Use of medication, except for oral blood glucose lowering medication
* Use of insulin
* All co-morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthritis, spasticity/rigidity, all neurological disorders and paralysis).
* HbA1c > 10.0% (86 mmol/mol)
* Donated blood in last 3 months
* Diagnosed impaired renal or liver function
* Myocardial infarction within the last 3 years
* Gastric acid inhibitors
* Use of anti-coagulants

Ages: 70 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Muscle protein fractional synthetic rate | -2, 0, +2, +5 h during the trial
  Muscle protein fractional synthetic rate assessed using the muscle biopsy technique.

SECONDARY OUTCOMES:
Plasma amino acids | every 30 min (from -2 h to + 5 h during the test day)
  Blood sampling will occur through a catheter placed in an anticubital vein every 30 minutes throughout the test day. We will be using this plasma to measure plasma amino acids to determine the enrichment of labeled amino acids from both the IV tracer and the intrinsically-labeled casein protein. We wish to track the changes in amino acids from the intrinsically-labeled casein protein.
Plasma nitrate | every 30 min (from -2 h to + 5 h during the test day)
  Plasma nitrate will be measured every 30 minutes during the test day through blood sampling from the catheter inserted into an antecubital vein. We want to measure the changes in plasma nitrate after consuming the nitrate or placebo beverage.

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Study Director — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356
- [Derived] Kouw IW, Gorissen SH, Burd NA, Cermak NM, Gijsen AP, van Kranenburg J, van Loon LJ. Postprandial Protein Handling Is Not Impaired in Type 2 Diabetes Patients When Compared With Normoglycemic Controls. J Clin Endocrinol Metab. 2015 Aug;100(8):3103-11. doi: 10.1210/jc.2015-1234. Epub 2015 Jun 2. PMID 26037513